CLINICAL TRIAL: NCT01329536
Title: The Occurrence of the ApoE4 Allele in Agitated In-Patients With Late-Onset Alzheimer's Disease Compared to Age- and Gender-Matched, Non-Agitated In-Patients With Late-Onset Alzheimer's Disease
Brief Title: The Occurrence of the ApoE4 Allele in Agitated In-Patients With Late-Onset Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: AIHBG-1380-Agitation
Record Dates: First submitted 2011-01-11; First posted 2011-04-06 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-02

CONDITIONS: Alzheimer's Disease; Agitation
Keywords: Alzheimer's Disease; Agitation; Genetics; Apolipoprotein; ApoE4
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva and blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- AD Patients with Agitation: Patients with a diagnosis of probable Alzheimer's Disease who show signs of agitation based on the Cohen-Mansfield Agitation Inventory
- AD Patients without Agitation: Patients with a diagnosis of probable Alzheimer's Disease who do not show signs of agitation based on the Cohen-Mansfield Agitation Inventory and are matched in both age and gender to the AD Patients with Agitation

SUMMARY:
The purpose of this clinical research study is to determine if a specific genetic allele is involved with the development of agitation in patients with late-onset Alzheimer's Disease (AD). The study will compare the results of genetic testing between two groups: individuals with late-onset AD who show signs of agitation and individuals with late-onset AD who do not show signs of agitation.

DETAILED DESCRIPTION:
Agitation and other behavioral disturbances are a main cause in the need for increasing levels of care for the patient with Alzheimer's disease (AD). And while the pathology of dementia has been studied in great detail, the etiology is considered multi-factorial. The hypothesis behind this clinical study is that the presence of the apo lipoprotein E4 (APO E4) allele will serve to predict which patients with late on-set AD are at greater risk to develop agitation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are at least 65 years of age
* Meet the DSM-IV-TR criteria for late-onset Alzheimer's Disease (AD)

Exclusion Criteria:

* Unable to provide informed consent or do not have a legally acceptable caregiver and/or representative present or available to enter into the informed consent process on the study subject's behalf
* Diagnosis of a non-Alzheimer's type of dementia
* Determined by the Principal Investigator (or his designee) that the study subject would be unsuitable for study participation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with a diagnosis of probable Alzheimer's Disease (late-onset)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Apolipoprotein E4 Allele | Single clinic visit (day 1)
  This study consists of a single clinic visit. After subject has completed the informed consent process and meets eligibility criteria, a blood sample and a saliva sample will be collected. Genetic results from this one-time specimen collection will be evaluated and compared with results from participants in the other study group of age- and gender-matched patients. Outcomes will be measured comparatively.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Reiners, MD, Principal Investigator — Avera McKennan Hospital & University Health Center
Locations (1):
- Avera Research Institute, Sioux Falls, South Dakota, United States

REFERENCES:
- [Background] Bynum JP, Rabins PV, Weller W, Niefeld M, Anderson GF, Wu AW. The relationship between a dementia diagnosis, chronic illness, medicare expenditures, and hospital use. J Am Geriatr Soc. 2004 Feb;52(2):187-94. doi: 10.1111/j.1532-5415.2004.52054.x. PMID 14728626
- [Background] Drachman DA. Aging of the brain, entropy, and Alzheimer disease. Neurology. 2006 Oct 24;67(8):1340-52. doi: 10.1212/01.wnl.0000240127.89601.83. PMID 17060558
- [Background] Mayeux R, Saunders AM, Shea S, Mirra S, Evans D, Roses AD, Hyman BT, Crain B, Tang MX, Phelps CH. Utility of the apolipoprotein E genotype in the diagnosis of Alzheimer's disease. Alzheimer's Disease Centers Consortium on Apolipoprotein E and Alzheimer's Disease. N Engl J Med. 1998 Feb 19;338(8):506-11. doi: 10.1056/NEJM199802193380804. PMID 9468467
- [Background] Mirakhur A, Craig D, Hart DJ, McLlroy SP, Passmore AP. Behavioural and psychological syndromes in Alzheimer's disease. Int J Geriatr Psychiatry. 2004 Nov;19(11):1035-9. doi: 10.1002/gps.1203. PMID 15481075
- [Background] Koss E, Weiner M, Ernesto C, Cohen-Mansfield J, Ferris SH, Grundman M, Schafer K, Sano M, Thal LJ, Thomas R, Whitehouse PJ. Assessing patterns of agitation in Alzheimer's disease patients with the Cohen-Mansfield Agitation Inventory. The Alzheimer's Disease Cooperative Study. Alzheimer Dis Assoc Disord. 1997;11 Suppl 2:S45-50. doi: 10.1097/00002093-199700112-00007. PMID 9236952
- [Background] Fitzpatrick AL, Kuller LH, Lopez OL, Kawas CH, Jagust W. Survival following dementia onset: Alzheimer's disease and vascular dementia. J Neurol Sci. 2005 Mar 15;229-230:43-9. doi: 10.1016/j.jns.2004.11.022. Epub 2004 Dec 23. PMID 15760618